CLINICAL TRIAL: NCT01892059
Title: A Randomized Controlled Trial Comparing the Segmental Artery Clamping and Main Renal Artery Clamping During Laparoscopic Partial Nephrectomy
Brief Title: Study of Segmental Renal Artery Clamping During Laparoscopic Partial Nephrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Changjun Yin, Head of Urology Department, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChiCTR-TRC-13003054
Record Dates: First submitted 2013-06-30; First posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-06

CONDITIONS: Kidney Neoplasms; Renal Cell Carcinoma
Keywords: renal tumour; partial nephrectomy; laparoscope; segmental renal artery clamping
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Segmental artery clamping (Experimental): Patients with Renal tumor are randomized into this group,they will received laparoscopic partial nephrectomy. During operation, the technique of segmental renal artery clamping will performed.
  Interventions: Procedure: Segmental artery clamping
- Main renal artery clamping (Active Comparator): Patients with renal tumor are randomized into this group,they will received laparoscopic partial nephrectomy. During operation, the technique of traditional main renal artery clamping will be performed.
  Interventions: Procedure: Main renal artery clamping

INTERVENTIONS:
Procedure: Segmental artery clamping — Laparoscopic partial nephrectomy with segmental artery clamping will be performed for patients enrolled in this group.
  Arms: Segmental artery clamping
Procedure: Main renal artery clamping — Laparoscopic partial nephrectomy with main renal artery clamping technique will be performed for patients enrolled in this group.
  Arms: Main renal artery clamping

SUMMARY:
The purpose of this study is to compare the efficacy and safety of the segmental artery clamping and main renal artery clamping during laparoscopic partial nephrectomy

DETAILED DESCRIPTION:
Renal tumor patients,for whom laparoscopic partial nephrectomy is suitable, will be randomly divided into two groups,segmental artery clamping group and main artery clamping group. All procedures were performed by the same laparoscopic surgeon. Blood loss, operation time, warm ischemia time, complications and affected renal function before and after operation will be recorded and compared. The safety and efficiency of laparoscopic partial nephrectomy with segmental renal artery clamping will be evaluated in comparison with the conventional main renal artery clamping technique.

ELIGIBILITY:
Inclusion Criteria:

* 20<age<70yr
* Stage T1a
* Patients volunteered for this study and provided written informed consent

Exclusion Criteria:

* Bilateral renal tumor
* tumor of solitary kidney
* glomerulonephritis
* renal insufficiency
* GFR of invalid kidney less than 30ml/min
* presence of suspect metastasis
* serious systematic disease: severe coagulation disorders
* important organ insufficiency and severe psychological disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Glomerular Filtration Rate | 3 months postoperative

SECONDARY OUTCOMES:
warm ischemia time | during surgery

OTHER OUTCOMES:
estimated blood loss | during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Changjun Yin, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Department of Urology, First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Shao P, Tang L, Li P, Xu Y, Qin C, Cao Q, Ju X, Meng X, Lv Q, Li J, Zhang W, Yin C. Precise segmental renal artery clamping under the guidance of dual-source computed tomography angiography during laparoscopic partial nephrectomy. Eur Urol. 2012 Dec;62(6):1001-8. doi: 10.1016/j.eururo.2012.05.056. Epub 2012 Jun 7. PMID 22695243
- [Background] Shao P, Tang L, Li P, Xu Y, Qin C, Cao Q, Ju X, Meng X, Lv Q, Li J, Zhang W, Yin C. Application of a vasculature model and standardization of the renal hilar approach in laparoscopic partial nephrectomy for precise segmental artery clamping. Eur Urol. 2013 Jun;63(6):1072-81. doi: 10.1016/j.eururo.2012.10.017. Epub 2012 Oct 24. PMID 23116655
- [Result] Shao P, Qin C, Yin C, Meng X, Ju X, Li J, Lv Q, Zhang W, Xu Z. Laparoscopic partial nephrectomy with segmental renal artery clamping: technique and clinical outcomes. Eur Urol. 2011 May;59(5):849-55. doi: 10.1016/j.eururo.2010.11.037. Epub 2010 Dec 7. PMID 21146917